CLINICAL TRIAL: NCT02129114
Title: A Multi-Center,Randomized,Non-Inferiority and Positively Controlled Clinical Trial to Evaluate the Safety and Efficacy of Dural Repair Patch in Neurosurgical Repairs
Brief Title: Study to Evaluate the Safety and Efficacy of Dural Repair Patch in Neurosurgical Repairs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medprin Regenerative Medical Technologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-CT-RK2014
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Neurosurgical Repairs

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReDura Onlay (Experimental): The Dural Repair Patch manufactured by Guangzhou Medprin Regenerative Medical Technologies Co., Ltd.
  Interventions: Device: ReDura Onlay
- DuraGen (Active Comparator): Dural Graft Matrix manufactured by Integra LifeSciences (U.S.) Corporation.
  Interventions: Device: DuraGen

INTERVENTIONS:
Device: ReDura Onlay — Subject will be clinically followed post-surgery until hospital discharge or within ten (10) days of the procedure and at three (3) months and six (6) months. The data up to and including the 6 month follow-up visit will be used in demonstrating the performance of ReDura Onlay.
  Arms: ReDura Onlay
Device: DuraGen — Subject will be clinically followed post-surgery until hospital discharge or within ten (10) days of the procedure and at three (3) months and six (6) months. The data up to and including the 6 month follow-up visit will be used in demonstrating the performance of DuraGen.
  Arms: DuraGen

SUMMARY:
1. Most of dural defects may lead to subcutaneous effusion and Cerebral Spinal Fluid (CSF) leakage, which may result in infection; besides, direct adhesion of brain tissues with sub-scalp tissues also increase the risk of epilepsy, in severe cases, dural defect is considered a life-threatening condition. So, it's important to repair the dura mater for restoring its full integrity .
2. Dural Repair Patch(ReDura Onlay) manufactured by Guangzhou Medprin Regenerative Medical Technologies Co., Ltd. As a product made of clinical absorbable polymer materials by using bionic technology, Dural Repair Patch has highly bionic 3-dimensional structure which is proved to facilitate migration and growth of regenerative cells, as well as to accelerate the growth and repairing of regenerative meninges. While the material is degraded gradually and absorbed by the body, regenerative meningeal tissue is gradually formed, achieving true reconstruction of the dura mater.
3. To evaluate the safety and effectiveness of Dural Repair Patch in neurosurgical repairs of dural defects.

DETAILED DESCRIPTION:
1. Dura mater is an important structural cell layer on the surface of brain serving as an important barrier for brain protection. Dural defects could be caused by a vast variety of factors, including trauma, tumor invasion, increased volume of the intra-cranial contents, certain congenital diseases, surgical procedures and etc. Most of dural defects may lead to subcutaneous effusion and CSF leakage, which may result in infection; besides, direct adhesion of brain tissues with sub-scalp tissues also increase the risk of epilepsy, in severe cases, dural defect is considered a life-threatening condition. Repairing of dura mater to restore its full integrity is proved to reduce the incidences of its complications, such as CSF leakage, epilepsy and etc. In particular, the outcomes of neurosurgeries are largely dependent of the post-operative integrity of dura mater.
2. most of the currently available products require surgical dural suturing, which elongate the duration of operation; nevertheless, some surgical site are unsuitable for suturing. The currently marketed non-suture dural substitutes and mainly made of a single material with a single-layered structure, which are significantly different from the natural structure of extracellular matrix, poorly mimicking the microstructure of dural mater; hence, the structures and surface properties of such products do not meet the requirements for local cellular regeneration post dural repairs, resulting in poor repair outcomes. Besides, the increased contractility of these products after water absorption also impose a certain extent of risk in practical application, since dural repairing surgeries are mainly conducted on the defective site of soft cerebral tissues.
3. As a product prepared by using bionic technology, Dural Repair Patch manufactured by Guangzhou Medprin Regenerative Medical Technologies Co., Ltd. is able to mimic porous fiber biomimetic structure that facilitate the cellular growth on the stent. Through effective control over the bionic technology parameters, the diameter, aperture and porosity of the fiber are almost identical to the in vivo tissue structure, so as to improve the cellular adhesion and growth on the sten. Increased strength, suitable ductility and improved hydrophilicity all contribute to the excellent flexibility and adhesiveness of the finished product able to adhesive closely to the autologous tissues, meeting the clinical requirements. Being made of absorbable polymer materials widely accepted in clinical product, the product has a highly bionic 3-dimensional structure which is proved to facilitate migration and growth of regenerative cells, as well as to accelerate the growth and repairing of regenerative meninges. While the material is degraded gradually and absorbed by the body, regenerative meningeal tissue is gradually formed, achieving true reconstruction of the dura mater.
4. Design and methods

4.1 Subjects who meet the inclusion criteria are randomized in accordance with the admission time; routine blood test, liver and kidney function test, as well as cellular and humoral immunity test are conducted prior to the surgery.

4.2 Location, characteristics and size of the defects,as well as the conditions of surgical incision are all observed intra-operatively.

4.3 Dura mater membrane repairing surgeries are conducted by closely attaching either an appropriately-sized test product or reference product to the defected part of dura mater membrane, before the incision in the skull is closed by using a conventional approach.

4.4 The subjects'conditions are reviewed on Day 1, 3, 5, 7 and 10 post operations, respectively.

4.5 Lumbar puncture is conducted on Day 10±2 post operation based on the subject's conditions, in order to measure the intracranial pressure and test for cerebrospinal fluid leakage; routine blood, liver and kidney function, as well as cellular and humoral immunity are re-tested on Day 10±2 post operation and the values obtained are compared with the pre-operative baseline measurements and recorded, so as to evaluate the clinical significance; On Day 10±2 post operation, cerebrospinal fluid leakage or subcutaneous effusion are examined by CT scan and clinical examinations, so as to assess the relationship of such events to the test/reference product.

4.6 For subjects who received a re-operation in the same location or a second neurosurgery, the conditions of test product or reference product in the repairing site is observed, e.g. examine (combined with histological test) product adhesion with cerebral tissues and etc.

4.7 The subjects are asked to attend a return visit or a telephone follow-up session on Day 90±10 and 180±20 post operation.

ELIGIBILITY:
Inclusion Criteria:

1. male or female aged 18-65 years;
2. whose expected survival is not less than 12 months
3. Patients with dura mater defects which occurred in a variety of neurosurgeries (including traumatic brain injury, brain tumors, cerebrovascular disease, congenital neurological diseases, intra-spinal diseases and etc.) and required surgical repairing.
4. All the enrolled subjects should not present obvious pre-operative inflammation symptoms,
5. Written informed consents were obtained from all of the patients and/or their guardians.

Exclusion Criteria:

1. Patient who present severe visceral (heart, liver, kidney, circulation system or etc.) diseases.
2. Patient with unstable vital signs.
3. Pregnant or lactating women.
4. Patient who have a past history of serious allergy
5. Patient who have a past history of severe immunodeficiency disease.
6. Other undesirable conditions set by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Rate of successful prevention of CSF leakage | Day 10±2 post operation
  on Day 10±2 post operation, occurrence of CSF leakage is checked on both CT and clinical examination

SECONDARY OUTCOMES:
Healing of scalp incision | 6 month
  the healing of scalp incision is reviewed on Day 3, Day 5, Day7, Day 10, Month 3 and Month 6, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Yi Quan, professor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China